CLINICAL TRIAL: NCT07279181
Title: Comparative Assessment of Transvaginal Ultrasound, Hysterosonography, and MRI in Uterine Niche
Brief Title: TVS, SHG, and MRI in Uterine Niche
Status: Completed | Type: Observational
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GKLW-2024-044-A
Record Dates: First submitted 2025-11-16; First posted 2025-12-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Uterine Niche
Keywords: Uterine niche; MRI; Ultrasound; Hysterosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women diagnosed with uterine niche: Women diagnosed with uterine niche, all patients underwent ultrasound, hysterosonography, and thin-slice MRI before surgery, and hysteroscopic evaluation of the niche was completed during the operation.

SUMMARY:
Uterine niche is a defect formed by poor healing of the lower uterine myometrium after cesarean section, defined as a depression of at least 2mm in the uterine myometrium at the cesarean scar; it is associated with gynecological symptoms and even life-threatening pregnancy complications, so accurate imaging evaluation is crucial for diagnosis, symptom grading, and treatment planning. Currently, transvaginal ultrasound (TVS), saline hysterosonography (SHG), and magnetic resonance imaging (MRI) are commonly used for evaluation, but there are controversies about the consistency of their measurements and repeatability of results. This observational study, conducted at the International Peace Maternity and Child Health Hospital affiliated with Shanghai Jiao Tong University School of Medicine, included women diagnosed with uterine niche.

ELIGIBILITY:
Inclusion Criteria:

* Women (18-45 years) diagnosed with CSD at our center.
* Women having postmenstrual spotting after CS
* Signed informed consent.

Exclusion Criteria:

* Women who has a positive urine pregnancy test.
* Presence of an intrauterine device.
* With poor image quality from image will be excluded.
* Refuse to participate in this study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample size is the actual number included within the study time frame
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Detection rates of niches | Periprocedural
  Detection rates of niches

SECONDARY OUTCOMES:
Residual myometrial thickness | Periprocedural
  Residual myometrial thickness of niches measured by TVS, SHG and MRI
The differences in the detection of abnormal structures | Periprocedural
  The differences in the detection of abnormal structures

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Study Chair — The International Peace Maternity & Child Health Hospital
Locations (1):
- International Peace Maternity & Child Health Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Ask the principal investigator by email

REFERENCES:
- [Background] Araujo Santana Tavares M, Busoletto Tripode BG, Kozlowski Andreucci B, Bezerra Cirne E, Almeida Sathler Bretas E, Rios Torres L, Oliveira Pacheco E, S Torres U, D'Ippolito G. Isthmic uterine lesions: a comprehensive pictorial review of MRI features and management strategies. Abdom Radiol (NY). 2025 Dec;50(12):6076-6084. doi: 10.1007/s00261-025-05037-0. Epub 2025 Jun 7. PMID 40481886
- [Background] Donnez O. Cesarean scar defects: management of an iatrogenic pathology whose prevalence has dramatically increased. Fertil Steril. 2020 Apr;113(4):704-716. doi: 10.1016/j.fertnstert.2020.01.037. PMID 32228874
- [Background] Klein Meuleman SJM, Min N, Hehenkamp WJK, Post Uiterweer ED, Huirne JAF, de Leeuw RA. The definition, diagnosis, and symptoms of the uterine niche - A systematic review. Best Pract Res Clin Obstet Gynaecol. 2023 Aug;90:102390. doi: 10.1016/j.bpobgyn.2023.102390. Epub 2023 Jul 15. PMID 37506497